CLINICAL TRIAL: NCT06388473
Title: Implementation of a Web-based App for Screening in Men in a Malaysian Primary Care Setting
Acronym: iScreenMen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NMRR-20-2188-56086 IIR
Record Dates: First submitted 2024-04-07; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Men's Health Screening; Implementation; Web-based Application
Keywords: mass screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored implementation intervention (Experimental): The tailored implementation intervention comprised of six implementation strategies: 1) Involve executive boards, 2) Mandate change, 3) Provide education and training, 4) Identify and prepare champions, 5) The use of information and communication technology and 6) Audit and provide feedback.
  Interventions: Behavioral: Tailored implementation intervention

INTERVENTIONS:
Behavioral: Tailored implementation intervention — The tailored implementation intervention comprised of six implementation strategies: 1) Involve executive boards, 2) Mandate change, 3) Provide education and training, 4) Identify and prepare champions, 5) The use of information and communication technology and 6) Audit and provide feedback.
  Other Names: ScreenMen

SUMMARY:
The purpose of this study is to determine how to successfully implement ScreenMen in the primary care setting. ScreenMen is a mobile web-based app that has been developed to increase the uptake of screening in men. ScreenMen undertook a vigorous and systematic approach in its development. It was developed based on theories, evidence and needs of men. ScreenMen particularly target men in the age group of 20 to 50 years as this group of men usually do not attend any health screening. This research is necessary because ScreenMen has yet to be implemented in the primary care setting. The study will last about five months and your participation will be about five months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthcare providers that were involved in the clinic health screening program.
2. Patients who were aged 18 years and above were eligible to participate.

Exclusion Criteria:

1. Temporary healthcare providers (working in the clinic less than six months during the study period) and those who were away on leave.
2. Patients who did not understand Bahasa Malaysia, English or Mandarin, cognitively impaired, had an active psychiatric illness or were too ill.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Reach | Beginning of intervention
  Number of healthcare providers who attended the workshop / Number of healthcare providers who were invited to the workshop.
Reach | Through study completion, 5 months.
  The number of patients who accessed ScreenMen.
Adoption of ScreenMen using qualitative methods | 5 months into study
  Factors affecting the participation of healthcare providers in adopting ScreenMen in daily practice using qualitative interviews.
Implementation of ScreenMen using qualitative methods | 5 months into study
  Factors affecting the implementation of ScreenMen daily practice using qualitative interviews.
Maintenance of ScreenMen using qualitative methods | 5 months into study
  Intention to implement ScreenMen and factors influencing the decision using qualitative methods.

SECONDARY OUTCOMES:
Impact of COVID-19 on the clinic using qualitative methods | 5 months into study
  The clinic situation during the COVID-19 pandemic and how it affected daily practice using qualitative methods.

CONTACTS AND LOCATIONS:
Overall Officials: Chirk Jenn Ng, PhD, Principal Investigator — University of Malaya
Locations (1):
- Klinik Kesihatan Cheras Baru, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ooi CY, Ng CJ, Sales A, Teo CH. Pilot implementation study of a web-based men's health screening app in primary care during COVID-19: a mixed-methods approach. BMC Health Serv Res. 2024 Oct 11;24(1):1219. doi: 10.1186/s12913-024-11702-9. PMID 39394132